CLINICAL TRIAL: NCT05271396
Title: Respiratory Functions and Respiratory Muscle Strength in Patients With Temporomandibular Joint Dysfunction
Status: Completed | Type: Observational
Sponsor: Halic University (Other)
Responsible Party: Principal Investigator, Seda Saka, Director, Halic University
Other Study IDs: ssaka3
Record Dates: First submitted 2022-02-17; First posted 2022-03-09 (Actual); Last update posted 2022-03-09 (Actual); Status verified 2022-03

CONDITIONS: Temporomandibular Joint Dysfunction Syndrome
Keywords: Temporomandibular Joint Dysfunction Syndrome
MeSH Terms: conditions — Temporomandibular Joint Dysfunction Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Temporomandibular Joint Dysfunction Group: Being diagnosed with Temporomandibular Joint Dysfunction
  Interventions: Other: Clinical Assessment
- Healthy-matched Group: Being healthy according to WHO criteria
  Interventions: Other: Clinical Assessment

INTERVENTIONS:
Other: Clinical Assessment — The demographic information and clinical findings of the participants were recorded. Mandible movements evaluation with a digital caliper. The Visual Analogue Scale (VAS) to measure the severity of pain at rest and during activity. Cervical lordosis and shoulder posture assessment, Fonseca Anamnestic Index for TMD severity classification. Spirometric measurement to evaluate respiratory functions of all participants and intraoral pressure measurement to determine respiratory muscle strength.

SUMMARY:
In our study, it was aimed to evaluate respiratory functions and respiratory muscle strength in patients diagnosed with temporomandibular dysfunction (TMD) and to compare them with healthy individuals. The study was conducted with a total of 46 participants, 23 of whom were diagnosed with TMD and 23 healthy individuals, at Batman Training and Research Hospital between August 2021 and December 2021. In the evaluation, the demographic information and clinical findings of the participants were recorded. Mandible movements were evaluated with a digital caliper. For TMJ, the Visual Analogue Scale (VAS) was used to measure the severity of pain at rest and during activity. Cervical lordosis and shoulder posture assessment was done by distance measurement. Fonseca Anamnestic Index was used for TMD severity classification. Spirometric measurement was performed to evaluate respiratory functions of all participants and intraoral pressure measurement was performed to determine respiratory muscle strength. Statistical analyzes were performed using the IBM SPSS Statistics 26 program. Significance level was accepted as p<0.05.

DETAILED DESCRIPTION:
In our study, it was aimed to evaluate respiratory functions and respiratory muscle strength in patients diagnosed with temporomandibular dysfunction (TMD) and to compare them with healthy individuals. The study was conducted with a total of 46 participants, 23 of whom were diagnosed with TMD and 23 healthy individuals, at Batman Training and Research Hospital between August 2021 and December 2021. In the evaluation, the demographic information and clinical findings of the participants were recorded. Mandible movements were evaluated with a digital caliper. For TMJ, the Visual Analogue Scale (VAS) was used to measure the severity of pain at rest and during activity. Cervical lordosis and shoulder posture assessment was done by distance measurement. Fonseca Anamnestic Index was used for TMD severity classification. Spirometric measurement was performed to evaluate respiratory functions of all participants and intraoral pressure measurement was performed to determine respiratory muscle strength. Statistical analyzes were performed using the IBM SPSS Statistics 26 program. Significance level was accepted as p<0.05.

ELIGIBILITY:
Inclusion Criteria:

* Volunteer to participate in the study.
* To be diagnosed with TMD for the TMD group,
* To be healthy according to WHO definition for healthy matched group
* Being between the ages of 17-50.

Exclusion Criteria:

* Having any previous pulmonary disease.
* To have experienced a TMD problem due to trauma.
* Having covid-19 in the last 6 months.

Ages: 17 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: The population of the study consists of cases diagnosed with TMD in Batman Training and Research Hospital between August 2021 and December 2021 and individuals who comply with the World Health Organization (WHO) definition of healthy person. The sample size of the study was calculated using the G-Power 3.1 (G-Power, Germany) program. The sample size was found to be 23 individuals in each group and a total of 46 individuals, with effect size 0.75, alpha 5%, and test power 80%.
Sampling Method: Probability Sample
Enrollment: 46 (Actual)
Dates: Start 2021-08-06 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2022-02-11 (Actual)

PRIMARY OUTCOMES:
FEV1 (liter) | at the enrollment
  This is the amount of air with pulmonary function test that the patient can force out of their lungs in one second.
FEV1 (%-percentage) | at the enrollment
  This is the percentage of air with pulmonary function test that the patient can force out of their lungs in one second.
FVC (liter) | at the enrollment
  This is the greatest total amount of air patient can forcefully breathe out after breathing in as deeply as possible.
FEV1/FVC (percentage) | at the enrollment
  The FEV1/FVC ratio is a number that represents the percentage of patient lung capacity patient is able to exhale in one second.
Inspiratory muscle test | at the enrollment
  Maximal inspiratory pressure (MIP) is going to measured using a mouth pressure meter (MicroRPM; MicroMedical, UK) according to the guideline of ATS and European Respiratory Society (ERS).
Expiratory muscle test | at the enrollment
  Maximal expiratory pressure (MEP) is going to measured using a mouth pressure meter (MicroRPM; MicroMedical, UK) according to the guideline of ATS and European Respiratory Society (ERS).

SECONDARY OUTCOMES:
Evaluation of Mandible Movements | at the enrollment
  Maximum mouth opening was evaluated with a digital caliper. In the measurement of maximum mouth opening, the patient was asked to open his mouth as wide as possible. The distance between the cutting edge of the upper incisor and the cutting edge of the lower incisor was measured in mm.
Cervical Lordosis and Shoulder Posture Evaluation | at the enrollment
  Auxiliary tools such as double-tri square, caliper, tape measure and ruler were used for distance measurements. While the patient was standing, the wall behind was taken as a reference, and the wall-acromion, wall-tragus, tragus-acromion and chin sternal notch were measured in centimeters (cm) in free posture. Participants were asked to look straight ahead, in the free posture used in daily life, their heels against the wall, their feet open at hip level. Measurements were made on the right and left sides with the help of ruler and tape measure.
Pain assessment | at the enrollment
  The Visual Analogue Scale (VAS) was used to evaluate the pain intensity of the participants at rest and during activity for the temporomandibular joint. The participants were told what the meaning of the number values between 0 and 10 on the horizontal chart, divided into 10 equal parts of 100 mm. "No pain" was 0 points, "Unbearable pain" was 10 points, "Moderate pain" was 5 points. Participants were asked to mark one of the values in line with these explanations and the values were recorded.
Temporomandibular joint dysfunction classification (Fonseca Index) | at the enrollment
  Fonseca Index consists of 10 questions. Participants were asked to answer each question. The scoring method was calculated as 'Yes (10 points)', 'Sometimes (5 points)' and 'No (0 points)'.
  Classification; TMD-No (0-15 points), Mild-TMD (20-45 points), Moderate-TMD (50-65 points), and Severe-TMD (70-100 points)

CONTACTS AND LOCATIONS:
Locations (1):
- Haliç University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided